CLINICAL TRIAL: NCT02351661
Title: The Nutrition Care In Canadian Hospitals Study: 2010-2013
Brief Title: The Nutrition Care in Canadian Hospitals Study; 2010-2013.
Acronym: CMTF
Status: Completed | Type: Observational
Sponsor: Canadian Malnutrition Task Force (Other)
Collaborators: Canadian Nutrition Society (Other)
Responsible Party: Principal Investigator, Heather Keller, Chair, Canadian Malnutrition Task Force
Other Study IDs: CMTF Prevalence 2010-2013
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- medica/surgical: Medical or surgical patients from 18 hospitals
  Interventions: Other: There was no intervention

INTERVENTIONS:
Other: There was no intervention — observational study, no intervention

SUMMARY:
The Nutrition Care In Canadian Hospitals study, conducted by the Canadian Malnutrition Task Force had the primary purpose of determining the prevalence of malnutrition in Canadian acute care hospitals. Secondary objectives were to determine the independent association of malnutrition with patient centred outcomes (e.g. length of stay) and describe the nutrition care processes for malnourished and well nourished patients.

DETAILED DESCRIPTION:
Data from 18 community and academic hospitals was collected from a convenience sample of 1022 medical or surgical patients. This prospective cohort study followed patients throughout their admission to 30-day post discharge. Measures included nutrition indicators, nutrition care processes and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* acute care admission, medical or surgical unit; English or French language;anticipated to stay in hospital for 2 or more days; consent to study entry;

Exclusion Criteria: other hospital units; palliative patients; unable to complete informed consent due to language barrier or no proxy available; dementia

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: medical or surgical patients; large hospitals (>250 beds) recruited 60 patients and small hospitals recruited 40 patients over the age of 18 years; all provided informed consent or proxy provided informed consent
Sampling Method: Non-Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
length of stay | 0- 60 days
  length of stay in acute care bed

CONTACTS AND LOCATIONS:
Overall Officials: Heather Keller, Principal Investigator — University of Waterloo

REFERENCES:
- [Background] Keller HH, Vesnaver E, Davidson B, Allard J, Laporte M, Bernier P, Payette H, Jeejeebhoy K, Duerksen D, Gramlich L. Providing quality nutrition care in acute care hospitals: perspectives of nutrition care personnel. J Hum Nutr Diet. 2014 Apr;27(2):192-202. doi: 10.1111/jhn.12170. Epub 2013 Oct 23. PMID 24147893
- [Result] Duerksen DR, Keller HH, Vesnaver E, Laporte M, Jeejeebhoy K, Payette H, Gramlich L, Bernier P, Allard JP. Nurses' Perceptions Regarding the Prevalence, Detection, and Causes of Malnutrition in Canadian Hospitals: Results of a Canadian Malnutrition Task Force Survey. JPEN J Parenter Enteral Nutr. 2016 Jan;40(1):100-6. doi: 10.1177/0148607114548227. Epub 2014 Sep 4. PMID 25189174
- [Result] Duerksen DR, Keller HH, Vesnaver E, Allard JP, Bernier P, Gramlich L, Payette H, Laporte M, Jeejeebhoy K. Physicians' perceptions regarding the detection and management of malnutrition in Canadian hospitals: results of a Canadian Malnutrition Task Force survey. JPEN J Parenter Enteral Nutr. 2015 May;39(4):410-7. doi: 10.1177/0148607114534731. Epub 2014 Jun 2. PMID 24894461
- [Derived] Jeejeebhoy KN, Keller H, Gramlich L, Allard JP, Laporte M, Duerksen DR, Payette H, Bernier P, Vesnaver E, Davidson B, Teterina A, Lou W. Nutritional assessment: comparison of clinical assessment and objective variables for the prediction of length of hospital stay and readmission. Am J Clin Nutr. 2015 May;101(5):956-65. doi: 10.3945/ajcn.114.098665. Epub 2015 Mar 4. PMID 25739926